CLINICAL TRIAL: NCT05149404
Title: The Application of Enhanced Recovery After Surgery Clinical Pathway in Posterior Cervical Spine Surgery:a Multicenter, Non-interventional Cohort Study
Brief Title: The Application of Enhanced Recovery After Surgery Clinical Pathway in Posterior Cervical Spine Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); Beijing Chao Yang Hospital (Other); Peking University International Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LM2020289
Record Dates: First submitted 2021-07-01; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-06

CONDITIONS: Cervical Spondylotic Myelopathy; Ossification of Posterior Longitudinal Ligament in Cervical Region
Keywords: enhanced recovery after surgery; Posterior cervical surgery; posterior cervical laminoplasty; Clinical pathway

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERAS group
- Conventional group

SUMMARY:
This study intends to establish a multidisciplinary collaborative ERAS clinical pathway of cervical posterior surgery,and to verify its effectiveness, safety and value in health economics.

DETAILED DESCRIPTION:
Enhanced recovery after surgery (ERAS) is a new model of deep cooperation between surgery，rehabilitation medicine, anesthesiology, nursing and other disciplines in recent years, which enables patients to start rehabilitation training as soon as possible after surgery and improves the comprehensive effect of surgery. Posterior cervical surgery is traumatic, and it is significant to enhance postoperative rehabilitation to improve the overall efficacy of patients. Currently, there are no clear guidelines supporting the clinical effectiveness of ERAS in reducing complications, reducing costs, and enhancing recovery after posterior cervical surgery. Therefore, this study aims to establish a multidisciplinary ERAS model for posterior cervical surgery in Peking University Third Hospital and verify its clinical effectiveness. This is a multi-center, multidisciplinary prospective cohort study,in which the orthopedics department was combined with the anesthesiology department, rehabilitation department, nutrition department, operating room and nursing team to establish the ERAS clinical pathways for posterior cervical spine surgery. Clinical pathways include surgical procedure optimization, rehabilitation procedure optimization, anesthesia and nursing procedure optimization. As it is optimized and promoted,the ERAS clinical pathways will improve the curative effect and prognosis of posterior cervical surgery, so that more patients with cervical spondylosis will benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70, gender unlimited;
2. Diagnostic diagnosis of cervical spondylosis and consistent with the indications of posterior spinal canal extended laminoplasty;
3. Basis of serious diseases of centerlessness, brain, lung, kidney or other important organs, preoperative ASA score I-II;
4. Agree to participate in the study and sign the informed consent.

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Preoperative ASA score ≥III;
  2. One-stage combined anterior and posterior surgery of cervical spine;
  3. Correction of cervical deformity;
  4. Patients with gastric emptied disorders (such as gastroesophageal reflux, chronic history of aspiration, delayed gastric emptied), complete obstruction of the digestive tract, and inability to use enteral preparations;
  5. Patients with high risk conditions, such as severe cardio-renal insufficiency, affecting the safety evaluation of the trial;
  6. People with mental disorders, alcohol dependence or drug abuse history;
  7. women in the period of lactation and pregnancy;
  8. People with allergic constitution or previous allergies to a variety of drugs;
  9. Other researchers consider it inappropriate to participate in this study
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
range of motion on X - ray | preoperation
  range of motion the neck in extension and flexion on X - ray
range of motion on X - ray | intraoperation
  range of motion the neck in extension and flexion on X - ray
range of motion on X - ray | 72 hours after surgery
  range of motion the neck in extension and flexion on X - ray
range of motion on X - ray | 3 months after surgery
  range of motion the neck in extension and flexion on X - ray
range of motion on X - ray | 6 months after surgery
  range of motion the neck in extension and flexion on X - ray
Japanese Orthopaedic Association Cervical Myelopathy Evaluation Questionnaire（JOACMEQ） | preoperation
  A questionare to evaluate the severity of cervical spondylosis myelopathy
Japanese Orthopaedic Association Cervical Myelopathy Evaluation Questionnaire（JOACMEQ） | intraoperation
  A questionare to evaluate the severity of cervical spondylosis myelopathy
Japanese Orthopaedic Association Cervical Myelopathy Evaluation Questionnaire（JOACMEQ） | 72 hours after surgery
  A questionare to evaluate the severity of cervical spondylosis myelopathy
Japanese Orthopaedic Association Cervical Myelopathy Evaluation Questionnaire（JOACMEQ） | 3 months after surgery
  A questionare to evaluate the severity of cervical spondylosis myelopathy
Japanese Orthopaedic Association Cervical Myelopathy Evaluation Questionnaire（JOACMEQ） | 6 months after surgery
  A questionare to evaluate the severity of cervical spondylosis myelopathy
multi-cervical-unit system（MCU） | preoperation
  To locate the cervical responsible section
multi-cervical-unit system（MCU） | intraoperation
  To locate the cervical responsible section
multi-cervical-unit system（MCU） | 72 hours after surgery
  To locate the cervical responsible section
multi-cervical-unit system（MCU） | 3 months after surgery
  To locate the cervical responsible section
multi-cervical-unit system（MCU） | 6 months after surgery
  To locate the cervical responsible section

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China